CLINICAL TRIAL: NCT01239186
Title: Identification and Characterization of the Methylation Abnormalities on Whole Genome Among Infertile Men
Acronym: METHYLHOMME
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOR 08027
Record Dates: First submitted 2010-10-22; First posted 2010-11-11 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Oligospermia
Keywords: methylation; micro array; locus H19; male infertility
MeSH Terms: conditions — Oligospermia; Infertility, Male

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sample of sperm collected by automasturbation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oligozoospermia: infertile patients presenting a reduced sperm count (less than 20 Millions of spermatozoa/ml)
  Interventions: Other: methylation analyses on spermatozoa from infertile men

INTERVENTIONS:
Other: methylation analyses on spermatozoa from infertile men — microarray analysis(www.EPIGENOMICS.com)

SUMMARY:
This study will analyse the sperm global methylation status of 62 infertile men before assisted reproductive techniques. Some of these patients (20%) present hypomethylation of H19 locus. A global methylation analysis may reveal others imprinting defects.

DETAILED DESCRIPTION:
An increase of the abnormalities of the imprint was brought back at the child's stemming from assisted reproductive techniques. Now abnormalities of methylation could be implied in defects of spermatogenesis and certain abnormalities of development of the male germ cells could be due to modifications abnormal epigenetics.

The objective of this research is to determine the frequency of arisen the abnormalities of methylation at the level of the locus H19 in the sperm cells of barren men presenting an unexplained oligozoospermia and to determine if these changes are a reflection of abnormalities of the profiles of methylation of the whole genome.

The patients will realize a taking of sperm having signed the consent.

ELIGIBILITY:
Inclusion Criteria:

* Men from 18 to 45 years old, presenting an idiopathic oligozoospermia lower than 10 million sperm cells / ml and include in a program of medically assisted conception
* Patients with social security
* Patients having signed the informed consent

Exclusion Criteria:

* Infertility with a neoplastic origin: patients subjected to a treatment potentially sterilizing (chemotherapy or radiotherapy).
* Infertility with an infectious origin
* Infertility with a traumatic origin
* Infertility bound to a chromosomal abnormality or a microdeletion of Y
* Histories of cryptorchidism, of varicocele

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Men from 18 to 45 years old, presenting an idiopathic oligozoospermia lower than 10 million sperm cells / ml and include in a program of medically assisted conception
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Bring to light methylation abnormalities of the locus H19 in men's mature sperm cells presenting an unexplained oligozoospermia | 1 day

SECONDARY OUTCOMES:
Determine if these methylation abnormalities of the locus H19 reflect changes in the profile of global methylation of the spermatic DNA | 1 day
Estimate the association between these modifications and the nuclear quality of the sperm cell | 1 day
  by TUNEL analysis
Estimate the association between these modifications and the rates of success with In VITRO fertilization | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Célia Ravel, MD, Principal Investigator — TENON Hospital - APHP
Locations (1):
- Department of Biology of reproduction (TENON Hospital), Paris, Île-de-France Region, France

REFERENCES:
- [Background] Adami HO, Bergstrom R, Mohner M, Zatonski W, Storm H, Ekbom A, Tretli S, Teppo L, Ziegler H, Rahu M, et al. Testicular cancer in nine northern European countries. Int J Cancer. 1994 Oct 1;59(1):33-8. doi: 10.1002/ijc.2910590108. PMID 7927900
- [Background] Anway MD, Cupp AS, Uzumcu M, Skinner MK. Epigenetic transgenerational actions of endocrine disruptors and male fertility. Science. 2005 Jun 3;308(5727):1466-9. doi: 10.1126/science.1108190. PMID 15933200
- [Background] Auger J, Kunstmann JM, Czyglik F, Jouannet P. Decline in semen quality among fertile men in Paris during the past 20 years. N Engl J Med. 1995 Feb 2;332(5):281-5. doi: 10.1056/NEJM199502023320501. PMID 7816062
- [Background] Carlsen E, Giwercman A, Keiding N, Skakkebaek NE. Evidence for decreasing quality of semen during past 50 years. BMJ. 1992 Sep 12;305(6854):609-13. doi: 10.1136/bmj.305.6854.609. PMID 1393072
- [Background] Davis TL, Yang GJ, McCarrey JR, Bartolomei MS. The H19 methylation imprint is erased and re-established differentially on the parental alleles during male germ cell development. Hum Mol Genet. 2000 Nov 22;9(19):2885-94. doi: 10.1093/hmg/9.19.2885. PMID 11092765
- [Background] Gicquel C, Gaston V, Mandelbaum J, Siffroi JP, Flahault A, Le Bouc Y. In vitro fertilization may increase the risk of Beckwith-Wiedemann syndrome related to the abnormal imprinting of the KCN1OT gene. Am J Hum Genet. 2003 May;72(5):1338-41. doi: 10.1086/374824. No abstract available. PMID 12772698
- [Background] Hartmann S, Bergmann M, Bohle RM, Weidner W, Steger K. Genetic imprinting during impaired spermatogenesis. Mol Hum Reprod. 2006 Jun;12(6):407-11. doi: 10.1093/molehr/gal040. Epub 2006 Apr 11. PMID 16608903
- [Background] Kaiser J. Developmental biology. Endocrine disrupters trigger fertility problems in multiple generations. Science. 2005 Jun 3;308(5727):1391-2. doi: 10.1126/science.308.5727.1391a. No abstract available. PMID 15933166
- [Background] Kobayashi H, Sato A, Otsu E, Hiura H, Tomatsu C, Utsunomiya T, Sasaki H, Yaegashi N, Arima T. Aberrant DNA methylation of imprinted loci in sperm from oligospermic patients. Hum Mol Genet. 2007 Nov 1;16(21):2542-51. doi: 10.1093/hmg/ddm187. Epub 2007 Jul 17. PMID 17636251
- [Background] Paulozzi LJ, Erickson JD, Jackson RJ. Hypospadias trends in two US surveillance systems. Pediatrics. 1997 Nov;100(5):831-4. doi: 10.1542/peds.100.5.831. PMID 9346983
- [Background] Preiksa RT, Zilaitiene B, Matulevicius V, Skakkebaek NE, Petersen JH, Jorgensen N, Toppari J. Higher than expected prevalence of congenital cryptorchidism in Lithuania: a study of 1204 boys at birth and 1 year follow-up. Hum Reprod. 2005 Jul;20(7):1928-32. doi: 10.1093/humrep/deh887. Epub 2005 Apr 28. PMID 15860495
- [Background] Skakkebaek NE, Rajpert-De Meyts E, Main KM. Testicular dysgenesis syndrome: an increasingly common developmental disorder with environmental aspects. Hum Reprod. 2001 May;16(5):972-8. doi: 10.1093/humrep/16.5.972. PMID 11331648
- [Background] Toppari J, Larsen JC, Christiansen P, Giwercman A, Grandjean P, Guillette LJ Jr, Jegou B, Jensen TK, Jouannet P, Keiding N, Leffers H, McLachlan JA, Meyer O, Muller J, Rajpert-De Meyts E, Scheike T, Sharpe R, Sumpter J, Skakkebaek NE. Male reproductive health and environmental xenoestrogens. Environ Health Perspect. 1996 Aug;104 Suppl 4(Suppl 4):741-803. doi: 10.1289/ehp.96104s4741. PMID 8880001